CLINICAL TRIAL: NCT03809234
Title: Effects of Pgp Transporter Inhibition on CNS Biodistribution of Ondansetron in Healthy Volunteers
Brief Title: Pgp Transporter and CNS Biodistribution of Ondansetron in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adverse effects related to study procedure (not study drug)
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Assistant Professor of Anesthsiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201811167
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Ondansetron; Sodium Chloride; tariquidar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ondansetron with Tariquidar (Experimental): The participants will receive an IV ondansetron infusion with tariquidar. Participants will receive either 8mg or 16 mg of iv ondansetron, with 4mg/kg tariguidar.
  Interventions: Drug: Ondansetron 8mg with Saline & Tariquidar; Drug: Ondansetron 16mg with Saline & Tariquidar
- Ondansetron with Placebo (Placebo Comparator): The participants will receive an IV ondansetron infusion with D5W as placebo. Participants will receive either 8mg or 16 mg of iv ondansetron.
  Interventions: Drug: Ondansetron 8mg with Saline & Tariquidar; Drug: Ondansetron 16mg with Saline & Tariquidar

INTERVENTIONS:
Drug: Ondansetron 8mg with Saline & Tariquidar — Each participant will receive two IV infusions of ondansetron, 24 hours apart. In the first and second sessions, respectively, placebo (D5W) or tariquidar (4mg/kg dose in D5W) 22 will be administered IV over 60 minutes. Ondansetron will be diluted in 50mL 0.9% normal saline, and tariquidar will be diluted in 250mL D5W.
Drug: Ondansetron 16mg with Saline & Tariquidar — Each participant will receive two IV infusions of ondansetron, 24 hours apart. In the first and second sessions, respectively, placebo (D5W) or tariquidar (4mg/kg dose in D5W) 22 will be administered IV over 60 minutes. Ondansetron will be diluted in 50mL 0.9% normal saline, and tariquidar will be diluted in 250mL D5W.

SUMMARY:
To determine the time-course of plasma and CSF concentrations of intravenous (IV) ondansetron in healthy subjects, with and without selective inhibition of Pgp efflux transporter.

DETAILED DESCRIPTION:
The study hypothesis is that inhibition of Pgp efflux transporters will increase the CNS bio-distribution of the 5-HT3R antagonist ondansetron.

Specifically:

1. Intravenous administration of ondansetron is expected to yield low CSF exposure.
2. Co-administration of ondansetron with intravenous tariquidar, an inhibitor of Pgp efflux transporters, will result in increased CSF exposure of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50;
2. Body mass index between 18.5 and 30;
3. Good general health with no remarkable medical conditions;
4. Able and willing to provide informed consent.

Exclusion Criteria:

1. Current pregnancy or lactation;
2. Known history of hepatic, renal, or cardiac disease, including Long QT Syndrome, cardiac arrhythmias or QTc interval >450msec;
3. Known hypertension, endocrine disorders (such as diabetes mellitus), chronic pain, hematologic disorders, or psychiatric conditions requiring medications;
4. Abnormal vital signs at screening visit, including:

   * HR <40 or >100
   * SBP < 90mmHg or >150mmHg
   * DBP > 100mmHg
5. Abnormal troponin values at screening visit
6. Abnormal complete blood count (CBC) or comprehensive metabolic panel (CMP) values at screening visit that could affect drug pharmacokinetics, or suggest undiagnosed medical condition which would increase the risk of complications resulting from this study.
7. Any contraindication for ondansetron administration;
8. Peri- or post-menopausal women experiencing symptoms such as hot flashes;
9. Contraindication to intrathecal catheter placement, such as known coagulopathy or history of clotting disorders, history of scoliosis or lumbar fusion, current infection or fever;
10. Ongoing use of any of the following medications with known effects on Pgp function: carbamazepine, phenytoin, phenobarbital, cyclosporine, clarithromycin, erythromycin, ritonavir, verapamil, rifampicin, St. John's wort;
11. Current treatment (or treatment within < 5 half-lives) with any medication, including QT-prolonging drugs and drugs known to have a significant interaction with ondansetron or P-gp substrates (see below:)

    * Antiretrovirals of Protease inhibitor (e.g. Ritonavir, Saquinavir) or Non-nucleoside reverse transcriptase inhibitors (e.g. Efavirenz, Zidovudine) family.
    * Phenytoin, Carbamazepine, Oxcarbazepine, Rifampin
    * Amiodarone
    * Azole antifungals (e.g. Itraconazole, Fluconazole)
    * Macrolide antibiotics (Erythromycin, Clarithromycin)
    * Cimetidine
    * Non-DHP calcium channel blockers Verapamil and Diltiazem
    * First generation antipsychotic medications Thioridazine, Haloperidol, Chlorpromazine, and Pimozide
    * Second generation antipsychotic medications Ziprasidone and Quetiapine
    * Antihistamine Terfenadine
    * Antidepressants Trazodone, Bupropion, monoamine oxidase inhibitors, Mirtazapine
    * Antiarrhythmics Propafenone, Flecainide, and Procainamide
    * Fluoroquinolone antibiotics Norfloxacin, Ofloxacin, and Ciprofloxacin
    * Cisapride
    * Fentanyl, Lithium, Tramadol
    * Intravenous Methylene blue
    * Other strong inhibitors or inducers of Cytochromes P450 2D6 or 3A4.
    * Other strong inhibitors or inducers of P-glycoprotein

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
CSF penetration of ondansetron with and without tariquidar - area under the curve (AUC) | 48 hours
  CSF penetration of intravenous ondansetron will be determined as AUCCSF0-∞ of ondansetron, and compared between the two sessions, with and without tariquidar

SECONDARY OUTCOMES:
Cmax CSF | 48 hours
  Maximum CSF concentration (Cmax CSF) of ondansetron, compared between the sessions
CSF:plasma concentration ratio | 48 hours
  CSF:plasma concentration ratio of ondansetron, compared between the two sessions
Plasma Cmax | 48 hours
  Maximum plasma concentration (Cmax) of ondansetron, compared between the sessions

OTHER OUTCOMES:
Evaluation of analgesic effect of ondansetron in an experimental heat pain model | 48 hours
  Comparison of analgesic effect of ondansetron in an experimental heat pain model: HPTT (as Δ°C from baseline) will be compared between the sessions at 30 min and 50 min after ondansetron infusion completion
Assessment of analgesic effect of ondansetron in an experimental cold pain model | 48 hours
  Comparison of analgesic effect of ondansetron in an experimental cold pain model duration of tolerance and pain rating after 120 second (or maximum tolerable) hand submersion in 3-5°C water will be compared between the sessions at 40 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Yawn BP, Wollan PC, Weingarten TN, Watson JC, Hooten WM, Melton LJ 3rd. The prevalence of neuropathic pain: clinical evaluation compared with screening tools in a community population. Pain Med. 2009 Apr;10(3):586-93. doi: 10.1111/j.1526-4637.2009.00588.x. Epub 2009 Mar 17. PMID 20849570
- [Background] Smith BH, Torrance N. Epidemiology of neuropathic pain and its impact on quality of life. Curr Pain Headache Rep. 2012 Jun;16(3):191-8. doi: 10.1007/s11916-012-0256-0. PMID 22395856
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Dogrul A, Ossipov MH, Porreca F. Differential mediation of descending pain facilitation and inhibition by spinal 5HT-3 and 5HT-7 receptors. Brain Res. 2009 Jul 14;1280:52-9. doi: 10.1016/j.brainres.2009.05.001. Epub 2009 May 8. PMID 19427839